CLINICAL TRIAL: NCT02891187
Title: Outpatient Visits Versus Telephone Interviews for Postoperative Care: A Randomized Controlled Trial
Brief Title: Visits Versus Telephone Calls for Postoperative Care
Acronym: OPTIONs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-103
Record Dates: First submitted 2016-08-10; First posted 2016-09-07 (Estimated); Results first posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-08

CONDITIONS: Satisfaction; Postoperative Complications; Pelvic Floor Disorder
Keywords: Postoperative Care; Telephone follow-up; Healthcare Value
MeSH Terms: conditions — Personal Satisfaction; Postoperative Complications; Pelvic Floor Disorders | interventions — Ambulatory Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Outpatient Clinic Visits (Active Comparator): Outpatient clinic visits for postoperative care is currently the standard of care. Patients who undergo surgery for a pelvic floor disorder will be scheduled appointments in the outpatient clinic at 1-2 weeks, 6 weeks, and 3 months where they will be evaluated by a physician.
  Interventions: Behavioral: Outpatient Clinic Visits
- Telephone Follow-up (Active Comparator): Patients will be called instead of returning to clinic for postoperative care at 1-2 weeks, 6 weeks, and 3 months.
  Interventions: Behavioral: Telephone follow-up

INTERVENTIONS:
Behavioral: Telephone follow-up — Patients will be called for postoperative care at 1-2 weeks, 6 weeks, and 3 months
  Arms: Telephone Follow-up
Behavioral: Outpatient Clinic Visits — Patients will return to the clinic at 1-2 weeks, 6 weeks, and 3 months
  Arms: Outpatient Clinic Visits

SUMMARY:
The OPTIONs study is a randomized controlled, non-inferiority study to evaluate postoperative care using outpatient clinic visits versus telephone calls for women undergoing surgery for pelvic floor disorders. The primary outcome is patient satisfaction using the Surgical-Consumer Assessment of Healthcare Providers and Systems (S-CAHPS) questionnaire provided by the Agency for Healthcare Research and Quality (AHRQ). Secondary outcomes include safety and cost analysis for patients' direct and indirect medical costs. Women who speak and understand either English or Spanish and planning to undergo an elective surgery for a pelvic disorder will be recruited. Baseline demographics, satisfaction, and cost analysis questionnaires will be acquired pre-operatively. Randomization will be assigned at the time of discharge from the hospital. Patients will either have scheduled clinic visits at 1-2 weeks, 6 weeks, and 3 months or telephone calls by a registered nurse at these same intervals. Questionnaires will be completed at 3 months for satisfaction and cost analysis.

DETAILED DESCRIPTION:
A. Objectives Healthcare in the United States is costly, does not result in high patient satisfaction and is in need of reform. It is well known that the current state of healthcare delivery is trapped in a paradox with higher spending and poorer outcomes compared to other countries. To bring American healthcare back on course, the focus must shift to value. Health care value relies on quality and cost with the following equation: value = quality ÷ cost. Quality incorporates clinical outcomes, safety, and patient satisfaction. Routinely, hospitals and providers are rated on their postoperative care using the Consumer Assessment of Healthcare Providers and Systems (S-CAHPS) endorsed by the Agency for Healthcare Research and Quality (AHRQ). (https://cahps.ahrq.gov) In this equation, value increases by improving quality with increasing patient satisfaction and/or lowering costs without negatively impacting outcomes and maintaining safety. All healthcare stakeholders including patients, payers, providers, and suppliers benefit from working towards improving value.

The value of routine, interval post-operative visits is unknown. Post-operative clinical visits are considered a "gold standard" based solely on tradition. Postoperative care of patients over the telephone has been utilized in place of traditional outpatient postoperative visits in the pediatric and adult surgery literature. Retrospectively, this form of postoperative care has proven to be safe, effective, and reduces patients' nonmedical costs with improvements in patient satisfaction as measured on non-validated global scales. However, a prospective trial evaluating patient satisfaction and the safety of phone call postoperative visits has not been undertaken. A key gap in assessing the value of Urogynecologic care is assessing the value of routine postoperative visits.

The specific aims for this study include the following:

1. Compare patient satisfaction with their postoperative care among women randomized to telephone calls versus routine outpatient visits at 3 months as measured by the postoperative domain of the S-CAHPS. Hypothesis: The investigators hypothesize that patients receiving postoperative care with telephone calls will report non-inferior satisfaction on the S-CAHPS as women who have in-person postoperative clinic visits.
2. Compare adverse events at 3 months between patients randomized to telephone calls versus postoperative visits. Hypothesis: The investigators hypothesize that adverse events will not differ between the two groups.
3. Determine the cost-effectiveness of postoperative care with telephone calls versus visits at 3 months using patient and societal perspectives. Hypothesis: The investigators hypothesize that postoperative care with phone calls is more cost-effective than in-person visits from both the patient and societal perspectives.

Ultimately, the long-term goal is to institute novel approaches to postoperative care that adds value to healthcare delivery. The overall objective is to replace routine postoperative visits with telephone follow-up in a non-inferiority randomized controlled trial of postoperative patients after surgery for a pelvic floor disorders. The central hypothesis is this novel use of telephone follow-up calls versus clinic visits in uncomplicated post-operative patients after surgery for pelvic floor disorders will result in non- inferior satisfaction for their care as well as significantly reduce patients' direct and indirect nonmedical costs for postoperative care. The hypothesis has been formulated on the basis of other retrospective, observational studies in the pediatric and adult surgery literature. The rationale for the proposed research is that, once it is established that postoperative care with telephone calls offers similar rates of satisfaction among patients for their postoperative care, that this new approach for healthcare will offer an alternative to routine postoperative care.

B. Study Design The investigators will conduct a randomized non-inferiority trial to compare patient satisfaction between outpatient visits and telephone calls for post-operative care. The investigators will recruit women pre-operatively at the UNM Urogynecology clinic who are undergoing surgery for pelvic floor disorders including urinary and/or anal incontinence and/or pelvic organ prolapse and/or pelvic pain, and/or mesh exposure/complications. All women will give written informed consent. Patients will be randomized at the time of discharge to either telephone follow-up or outpatient visits. Computer generated randomization will be assigned by research staff uninvolved with recruitment and will be stored in opaque, sequentially numbered envelops. Follow-up for both randomization arms will be scheduled at 1-2 weeks, 6 weeks, and 3 months post-operatively, as these are common timeframes for routine postoperative visits in our practice.

C. Number of Subjects The recruitment goal for this study is 120 patients to allocate 60 patients in the clinic visit group and 60 patients in the telephone follow-up group.

The sample size for this study is determined by our primary objective, patient satisfaction measured by the Consumer Assessment of Healthcare Providers and Systems (S-CAHPS) survey. The investigators will conduct a non-inferiority patient satisfaction study comparing postoperative care with clinic visits versus telephone calls.

The investigators have been able to identify two publications that have used the S-CAHPS; both of these reported scores for individual items, as well as composites of "top box" responses for individual items. For example, responses for the question, "After your surgery did the surgeon listen carefully to you?" has three responses: 1. Yes, definitely, 2. Yes, somewhat, and 3. No. A top box response is "Yes, definitely". The global satisfaction with their surgeon is a single item, ranging from 0 (worst surgeon possible) to 100 (best surgeon possible), with "top" box responses of 100. "Top" box responses in prior studies ranged from 56-100% with the majority of responses about 90%. Assuming both the control and experimental groups are equivalent in patient satisfaction, a non-inferiority calculation can be applied using 90% as the percentage "success" in the control group and experimental groups with 80% power, an alpha of 0.05, and 15% non-inferiority limit. In this equation, if there is truly no difference between the control and experimental groups, then 100 patients for total sample size are required to be 80% sure that the upper limit of a 90% two-sided confidence interval will exclude a difference in favor of the control group of more than 15%. The primary outcome measure is the global composite for the surgeon rating, which has been used in the previous studies. This sample size will provide similar power for comparison of other items and scale of the S-CAHPS between groups. The investigators anticipate that up to 10% of women who are recruited will have complications that preclude them from participation after consent and prior to randomization, such as poorly controlled pain, complications or surgeon concerns. In addition, the investigators anticipate that 10% of women will be lost to follow-up. Therefore the plan is to recruit a total of 120 women, 60 per group.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≥ 18 years of age
2. Women undergoing surgery for a pelvic floor disorder
3. Able to give informed consent
4. Has a reliable phone number for contact postoperatively
5. Able to speak and understand English or Spanish. Spanish forms will be submitted after initial review of English materials.

Exclusion Criteria:

1. Any patient whose physician decides medical necessity for the patient to have postoperative follow-up in the clinic
2. Unable to give written informed consent
3. Does not have a reliable phone number
4. Inability to speak and understand either English or Spanish. As noted above, Spanish forms will be submitted after initial review of English materials.
5. Those who specifically request postoperative clinic visits
6. Pregnant patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca G Rogers, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico Health Sciences, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] Squires D, Anderson C. U.S. health care from a global perspective: spending, use of services, prices, and health in 13 countries. Issue Brief (Commonw Fund). 2015 Oct;15:1-15. PMID 26591905
- [Background] Cortese DA, Korsmo JO. Putting U.S. health care on the right track. N Engl J Med. 2009 Oct 1;361(14):1326-7. doi: 10.1056/NEJMp0907561. Epub 2009 Sep 23. No abstract available. PMID 19776399
- [Background] Porter ME. What is value in health care? N Engl J Med. 2010 Dec 23;363(26):2477-81. doi: 10.1056/NEJMp1011024. Epub 2010 Dec 8. No abstract available. PMID 21142528
- [Background] Fischer K, Hogan V, Jager A, von Allmen D. Efficacy and utility of phone call follow-up after pediatric general surgery versus traditional clinic follow-up. Perm J. 2015 Winter;19(1):11-4. doi: 10.7812/TPP/14-017. PMID 25663201
- [Background] Rosbe KW, Jones D, Jalisi S, Bray MA. Efficacy of postoperative follow-up telephone calls for patients who underwent adenotonsillectomy. Arch Otolaryngol Head Neck Surg. 2000 Jun;126(6):718-21; discussion 722. doi: 10.1001/archotol.126.6.718. PMID 10864107
- [Background] Kimman ML, Dirksen CD, Voogd AC, Falger P, Gijsen BC, Thuring M, Lenssen A, van der Ent F, Verkeyn J, Haekens C, Hupperets P, Nuytinck JK, van Riet Y, Brenninkmeijer SJ, Scheijmans LJ, Kessels A, Lambin P, Boersma LJ. Economic evaluation of four follow-up strategies after curative treatment for breast cancer: results of an RCT. Eur J Cancer. 2011 May;47(8):1175-85. doi: 10.1016/j.ejca.2010.12.017. Epub 2011 Jan 21. PMID 21257305
- [Background] Uppal S, Nadig S, Smith L, Coatesworth AP. A cost-effectiveness analysis of conventional and nurse-led telephone follow-up after nasal septal surgery. Ann R Coll Surg Engl. 2004 Jul;86(4):243-6. doi: 10.1308/147870804515. PMID 15239863
- [Background] Gray RT, Sut MK, Badger SA, Harvey CF. Post-operative telephone review is cost-effective and acceptable to patients. Ulster Med J. 2010 May;79(2):76-9. PMID 21116423
- [Background] Hwa K, Wren SM. Telehealth follow-up in lieu of postoperative clinic visit for ambulatory surgery: results of a pilot program. JAMA Surg. 2013 Sep;148(9):823-7. doi: 10.1001/jamasurg.2013.2672. PMID 23842982
- [Background] Fallaize RC, Tinline-Purvis C, Dixon AR, Pullyblank AM. Telephone follow-up following office anorectal surgery. Ann R Coll Surg Engl. 2008 Sep;90(6):464-6. doi: 10.1308/003588408X300975. Epub 2008 Jul 2. PMID 18598594
- [Derived] Thompson JC, Cichowski SB, Rogers RG, Qeadan F, Zambrano J, Wenzl C, Jeppson PC, Dunivan GC, Komesu YM. Outpatient visits versus telephone interviews for postoperative care: a randomized controlled trial. Int Urogynecol J. 2019 Oct;30(10):1639-1646. doi: 10.1007/s00192-019-03895-z. Epub 2019 Feb 19. PMID 30783704

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 patients withdrew from the study prior to randomization- surgery cancellations or surgeon preference for clinic follow-up.
Period: Overall Study
Arm/Group | Outpatient Clinic Visits | Telephone Follow-up
Started | 51 | 52
Completed | 50 | 50
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Outpatient Clinic Visits | Telephone Follow-up | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (12.0) | 57.9 (12.9) | 58.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 21 | 48
  Not Hispanic or Latino | 22 | 24 | 46
  Unknown or Not Reported | 1 | 5 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 10 | 13
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 31 | 29 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 11 | 27
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 50
Language [Count of Participants; unit: Participants]
  English | 42 | 44 | 86
  Spanish | 8 | 6 | 14
Marital Status [Count of Participants; unit: Participants]
  Single | 13 | 3 | 16
  Married/Partner | 23 | 30 | 53
  Divorced/Separated | 6 | 9 | 15
  Widowed | 8 | 8 | 16
Education [Count of Participants; unit: Participants]
  Less than high school | 7 | 8 | 15
  High school/GED | 14 | 20 | 34
  Associate College Degree | 17 | 12 | 29
  4 year College Degree | 6 | 4 | 10
  Graduate Degree | 5 | 5 | 10
  Unknown/Not reported | 1 | 1 | 2
Annual Income [Count of Participants; unit: Participants]
  <$25,000 | 22 | 23 | 45
  %25,000-49,999 | 10 | 13 | 23
  $50,000-74,999 | 5 | 7 | 12
  $75,000-99,999 | 5 | 1 | 6
  >$100,000 | 7 | 4 | 11
  Unknown | 1 | 2 | 3
Living Arrangements [Count of Participants; unit: Participants]
  Alone | 12 | 8 | 20
  With spouse or other | 25 | 33 | 58
  Unknown or Not reported | 13 | 9 | 22
Miles from surgical facility [Mean (Standard Deviation); unit: miles] | 73.2 (88) | 78.97 (87.1) | 76.1 (87.2)
type of surgery [Count of Participants; unit: Participants]
  outpatient surgery | 21 | 18 | 39
  inpatient surgery | 29 | 32 | 61

OUTCOME MEASURES:

1. Primary Outcome: Patient Satisfaction
Description: The objective is to compare patient satisfaction between women who present for clinic postoperative visits versus telephone follow-up. The investigators hypothesize that telephone calls will show non-inferior patient satisfaction when compared to clinic postoperative visits. The investigators will test the working hypothesis by using the approach of randomizing patients undergoing surgery for PFDs to either telephone follow-up or routine outpatient visits for their postoperative care and utilizing the S-CAHPS questionnaire preoperatively and 3 months postoperatively.
Time Frame: Preoperative until 3 months postoperative
Population: "top box" rating on teh S-CAHPS questionnaire
Measure: Number; unit: participants
Arm/Group | Outpatient Clinic Visits | Telephone Follow-up
Number analyzed (Participants) | 50 | 50
participants
  Information to help you prepare for surgery | 43 | 42
  How well surgeon communicates with patients before surgery | 43 | 45
  Surgeon's attentiveness on day of surgery | 40 | 44
  Information to help you recover from surgery | 37 | 39
  How well surgeon communicates with patients after surgery | 38 | 15
  Helpful, courteous, and respectful staff at surgeon's office | 46 | 46
  Rating of surgeon | 46 | 44

2. Secondary Outcome: Adverse Events
Description: The objective is to demonstrate telephone follow-up as both an effective and safe modality for postoperative care. The investigators hypothesize telephone calls and outpatient visits will not show a significant difference in adverse outcomes or patient outcomes for their pelvic floor dysfunction. Adverse events will be captured during the 3 months postoperative period for both groups in this study.
Time Frame: 3 months postoperative
Population: Adverse events included urinary tract infection, readmission, re-operation within 3 months, intraoperative complications, and other
Measure: Count of Participants; unit: Participants
Arm/Group | Outpatient Clinic Visits | Telephone Follow-up
Number analyzed (Participants) | 50 | 50
Participants | 15 | 11

ADVERSE EVENTS:
Time Frame: Adverse events were recorded 3 months postoperatively
Description: We used the definition provided by clinical trails
Arm/Group | Outpatient Clinic Visits | Telephone Follow-up
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/50 | 3/50
Other Adverse Events (participants affected / at risk) | 12/50 | 8/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Outpatient Clinic Visits (N=50) | Telephone Follow-up (N=50)
Readmission (Surgical and medical procedures) | 3 (3) | 3 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Outpatient Clinic Visits (N=50) | Telephone Follow-up (N=50)
Infection, other (Surgical and medical procedures) | 12 (12) | 8 (8) — Urinary tract infection and other outpatient infection management

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT02891187/Prot_SAP_000.pdf